CLINICAL TRIAL: NCT02208856
Title: Safety, Pharmacokinetics and Pharmacodynamics of Single Rising Doses (1, 4, 15, 50, 100, 200, 400, and 600 mg) Oral BIRB 796 BS in Healthy Human Subjects. A Placebo Controlled, Randomised Study, Double Blinded at Each Dose Level
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of Single Rising Doses Oral BIRB 796 BS in Healthy Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1175.1
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BIBR 796 BS food effect (Experimental)
  Interventions: Drug: BIBR 796 BS; Other: high fat standardized breakfast
- BIBR 796 BS (Experimental)
  Interventions: Drug: BIBR 796 BS

INTERVENTIONS:
Drug: BIBR 796 BS
  Arms: BIBR 796 BS; BIBR 796 BS food effect
Drug: Placebo
  Arms: Placebo
Other: high fat standardized breakfast
  Arms: BIBR 796 BS food effect

SUMMARY:
To assess safety, pharmacokinetics and pharmacodynamics of BIRB 796 BS in escalating single doses, with and without a 64 g fat breakfast at one selected dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with good clinical practice (GCP) and local legislation
* Age >= 18 and <= 45 years
* Broca >= -20% and <= +20%

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant ot the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) (= 1 month prior to administration or during the trial)
* Use of any drugs, which might influence the results of the trial (= 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (=2 months prior to administration or during trial)
* Smoker (> 10 cigarettes of > 3 cigars of > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation > 400 ml (=1 month prior to administration of during the trial)
* Excessive physical activities (= 5 days prior to administration or during the trial)
* Any laboratory value outside the reference range of clinical relevance (but not exclusive to) total white cell count >= 10 x 10**9/L, C-reactive protein >= 4.5 mg/L, any haemoglobin or > 15 mg/dl protein on urine dipstick
* History of any familial bleeding disorder

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 1999-09; Primary Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with clinically relevant changes in vital signs | Baseline, up to 96 hours after drug administration
Number of subjects with clinically relevant changes in laboratory measurements | Baseline, up to 96 hours after drug administration
Number of subjects with clinically relevant changes in electrocardiograms (ECG) | Baseline, up to 96 hours after drug administration
Number of subjects with adverse events | up to 96 hours after drug administration

SECONDARY OUTCOMES:
Maximum concentration of the analyte in plasma (Cmax) | up to 48 hours after drug administration
Area under the concentration-time curve of the analyte in plasma from time zero to infinity (AUC0-inf) | up to 48 hours after drug administration
Time from dosing to the maximum concentration of the analyte in plasma (Tmax) | up to 48 hours after drug administration
Terminal rate constant of the analyte in plasma (λz) | up to 48 hours after drug administration
Half life of the analyte in plasma (t1/2) | up to 48 hours after drug administration
Mean residence time of the analyte in the body (MRTtot) | up to 48 hours after drug administration
Apparent clearance of the analyte in plasma (CL/F) | up to 96 hours after drug administration
Apparent volume of distribution during the terminal phase λz (Vz/F) | up to 48 hours after drug administration
Mac-1/L selectin ratio of formyl-methionyl-leucyl-phenylalanine (fMLP)-stimulated to unstimulated neutrophils | up to 48 hours after drug administration
Mac-1/L selectin ratio of TNFalpha-stimulated to unstimulated neutrophils | up to 48 hours after drug administration
Percent changes in TNFalpha production | up to 48 hours after drug administration
  after ex vivo stimulation of whole blood with endotoxin